CLINICAL TRIAL: NCT06015555
Title: Effect Of Postural Control Exercise Versus¬¬ Tscharnuter Akademie For Motor Organization (TAMO) Therapy On Range Of Motion And Motor Function In Children With Congenital Muscular Torticollis
Brief Title: TAMO Therapy Versus Postural Control Exercise in Children With Congenital Muscular Torticollis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: khadija liaquat (Other)
Responsible Party: Sponsor-Investigator, khadija liaquat, Senior lecturer, Riphah International University
Organization: Riphah International University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU- Farhan
Record Dates: First submitted 2023-08-08; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Torticollis Congenital
MeSH Terms: conditions — Congenital torticollis | interventions — 14-thioglycolamido-7,8-dihydromorphinone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The TAMO therapy (Experimental): For four months, TAMO therapy will last 30 minutes every day, twice a week. The therapist first applies light loading for a short period of time to his left hemiocciput directed toward the supporting surface.
  Interventions: Behavioral: TAMO
- Postural Control exercises (Experimental): For four months, posture control exercises will be taught twice a week for 30 minutes each time. Under the age of 3 months, infants were required to shift their chin as far to the affected side and upward in the supine or dominant prone posture before they could regulate their neck. Instead of passively adjusting the newborns' heads, we waited for them to actively turn toward their midline.
  Interventions: Behavioral: Postural Control exercises

INTERVENTIONS:
Behavioral: TAMO — TAMO therapy
  Arms: The TAMO therapy
Behavioral: Postural Control exercises — Postural Control exercises
  Arms: Postural Control exercises

SUMMARY:
A randomized control trial was conducted through convenient sampling. 18 subjects were randomly allocated into two groups, group A received postural control exercises in addition to conventional therapy, while Group B received TAMO therapy along with conventional therapy. analysis.

DETAILED DESCRIPTION:
Torticollis is common in children and can be congenital or acquired. Acquired cases can result from neck muscles or bone injuries. Though distressing for parents, it usually improves over time. Treatment includes postural control exercise and TAMO therapy, along with conventional treatment. To compare the effects of TAMO therapy versus postural control exercises on children with congenital muscular torticollis on cervical range of motion. A randomized control trial was conducted through convenient sampling. Eighteen subjects were randomly allocated into two groups; Group A received postural control exercises in addition to conventional therapy, while group B received TAMO therapy along with conventional therapy. The duration of the treatment was eight weeks. Goniometer, still photography, muscle function. Eighteen participants (n=18) were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 3 months
* Both genders
* Abnormal neck posture
* Torticollis of both sides

Exclusion Criteria:

* SCM mass present
* Deficit in cervical PROM greater than 15 degree
* Craniosynostosis (it is a birth defect in which the bones in a baby skull join together too early)
* Infectious
* Metabolic
* Scoliosis of spine
* Developmental plagiocephaly
* SCM tumor
* Visual disorder

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Goniometer | Readings were taken at baseline and four months of intervention
  It measured cervical range of motion.
Muscle function Scale: | Readings were taken at baseline and four months of intervention
  MFS is a tool used to check the function of the lateral flexors, a scale of 0 to 5, with higher scores indicating better function of muscles.Readings were taken at baseline and after four months of intervention of the neck in children,

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah Rehabilitation Center, Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided